CLINICAL TRIAL: NCT06492369
Title: The Accuracy of MAFLD Fibrosis Score in Detecting Fibrotic NASH in MAFLD Egyptian Patients
Brief Title: MAFLD Fibrosis Score for Detecting Fibrotic NASH in MAFLD Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Principle Investigator, Tanta University
Other Study IDs: 36264PR614/3/24
Record Dates: First submitted 2024-06-12; First posted 2024-07-09 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Metabolic- Associated Fatty Liver Disease (MAFLD)
Keywords: Metabolic- associated fatty liver disease (MAFLD); Fibrotic NASH; MAFLD fibrosis score (MFS)

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Metabolic-associated fatty liver disease (MAFLD), is a metabolic stress-induced liver injury characterized by diffuse hepatocyte macrovesicular fatty infiltration.

The incidence of MAFLD is increasing yearly, and its incidence rate is as high as 20% to 30% on a global scale, which seriously affects people's health. Non-alcoholic steatohepatitis (NASH), a chronic hepatitis that can progress to advanced fibrosis, decompensated cirrhosis, and hepatocellular carcinoma, affects one-fifth of NAFLD patients. Depending on the histological severity of fibrosis, patients with NASH can be further classified as early NASH (F0-F1 fibrosis), fibrotic NASH (≥F2 fibrosis), or NASH-cirrhosis (F4 fibrosis).

Identifying subjects with fibrotic NASH is essential as they are at risk of complications, and disease progression and may benefit from potential pharmacological therapy.

Assessment of fibrotic NASH ranges from noninvasive scores to percutaneous liver biopsy, but liver biopsy is invasive and limited by cost, sampling variability, and intrareader/interreader variability.

Noninvasive modalities to risk stratify fibrotic NASH include serum biomarkers, imaging, and algorithms combining both. The FibroScan-AST (FAST) composite score is based on the liver stiffness measure (LSM), controlled attenuation potential (CAP), and AST. At the cut-off of a FAST score ≥0.67, biopsy-proven fibrotic NASH (NAFLD with a histological NAFLD activity score [NAS] ≥4 and fibrosis ≥2) can be ruled in with 90% specificity.

A new predictive model was recently developed based on eight variables (age, BMI, HbA1c, history of type 2 diabetes, International normalized ratio (INR), AST, Gamma Glutamyl transferase (GGT), and platelet count). A composite score MAFLD Fibrosis Score (MFS) was calculated as: MFS = 0.078 × Age (year)-0.007363 × Platelet count (109/L) + 0.0146 × AST (U/L) + 0.007618 × GGT (U/L) + 6.673 × INR + 0.09833 × BMI (kg/m2) + 1.425 × type 2 diabetes (yes = 1, no = 0).

So, in this study, the investigators will try to evaluate the accuracy of the new emerging predictor MAFLD Fibrosis Score (MFS) vs AST- to-platelet ratio index (APRI) score, fibrosis-4 index (FIB-4) score, and NAFLD fibrosis score in the assessment of the fibrotic NASH in Egyptian NAFLD patients.

DETAILED DESCRIPTION:
This study will be a cross-sectional study and will be carried out on 380 MAFLD patients attending to Tanta tropical medicine outpatient clinic, faculty of medicine. The start of the research will be in March 2024 to August 2024 or until collecting the cases.

Sample size The study will be carried on 382 patients according to the prevalence in Egypt 47.5% with confidence level 95% and margin of error 5 All the patients will be subjected to;

History taking:

Full history taking including:

* Personal history (name, age, sex, occupation, residence and marital state).
* Anthropometric measures: weight, length, BMI, Waist circumference.
* Complaint.

Investigations:

* Complete blood picture (CBC).
* Lipid profile (triglycerides, HDL, LDL, cholesterol level).
* Fasting Blood glucose level and or HBA1C.
* Liver functions (ALT, AST, INR, GGT, albumin, bilirubin).
* Viral markers and Anti-nuclear antibody (ANA). Data of radiological examination

  * Fibroscan: Liver fibrosis and steatosis can be staged using Dimensional ultrasound transient elastography (TE).
  * Ultrasound on abdomen and pelvis for evaluation of liver condition.
  * Fibrotic NASH was diagnosed with FAST score with a cut-off ≥0.67, biopsy-proven fibrotic NASH (NAFLD with a histological NAFLD activity score [NAS] ≥4 and fibrosis ≥2). [8]
  * MAFLD fibrosis score (MFS) is calculated using the formula:

MFS = 0.078 × Age (year)-0.007363 × Platelet count (109/L) + 0.0146 × AST (U/L) + 0.007618 × GGT (U/L) + 6.673 × INR + 0.09833 × BMI (kg/m2) + 1.425 × type 2 diabetes (yes = 1, no = 0).[9] - The FIB-4 index is calculated using the formula: FIB-4= Age (years)×AST(U/L)/ [platelet (109/L) ×ALT 1/2 (U/L)].

- NAFLD fibrosis score (NFS) is calculated using the formula: NFS = -1.675 + 0.037 × age (year) + 0.094 × BMI (kg/m2) + 1.13 × impaired fasting glucose (IFG)/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet count (×109/L) - 0.66 × albumin (g/dL).

Ethical considerations:

* A written informed consent form authorizing the collection of this data was signed by all patients.
* The study will be approved by the Ethical Committee of the Faculty of Medicine at Tanta University.

The risks to the participants and measures needed to minimize these risks:

* The privacy of the data of the patients will be maintained (the procedure will be discussed later in this protocol.
* Any unexpected risks appeared during the course of research will be cleared to the patients and the ethical committee on time.

Adequate provisions to maintain privacy of participants and confidentially of data are as follow:

* A code number for each patient will be used, symbols to the name and address will be kept in a special file.
* The investigators will hide the patients' names when the research is used.
* The investigators will use the results of the research only in scientific aim and not use it in other

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 years.
* NAFLD Patients assessed by ultrasound, fibroscan.

Exclusion Criteria:

* Patients aged < 18 years
* pregnant women.
* Excess alcohol intake (more than 30 g in men and 20 g in women).
* Viral hepatitis.
* Autoimmune hepatitis
* secondary fatty liver (e.g., the use of systemic steroids or methotrexate).
* history of malignancy in the past 2 years.
* Unwilling to participate in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NAFLD patients attending Tanta Tropical Medicine outpatient clinic, faculty of medicine.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of MFS in detecting Fibrotic NASH | till August 2024
  evaluation of accuracy of MAFLD Fibrosis Score (MFS) in the assessment of the fibrotic NASH in Egyptian patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Tanta University Hospitals, Tanta, Gharbyea, Egypt